CLINICAL TRIAL: NCT00170820
Title: A Single Arm, Prospective, Open-label, Pilot Study to Assess Effects of the Switch From Sirolimus to Everolimus in Stable Maintenance Renal Transplant Patients Receiving a Calcineurin Inhibitor Free Regimen
Brief Title: Efficacy and Safety of the Switch From Sirolimus to Everolimus in Stable Maintenance Renal Transplant Patients Receiving a Calcineurin Inhibitor Free Regimen
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CRAD001AFR04
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Renal Transplantation
Keywords: Renal transplantation, maintenance, switch, everolimus, CNI-free
MeSH Terms: interventions — Everolimus

INTERVENTIONS:
Drug: Everolimus

SUMMARY:
The purpose of this study is to assess if a combination of everolimus, steroids, and mycophenolate mofetil is associated with a better renal function than sirolimus.

ELIGIBILITY:
Inclusion Criteria:

* First or second renal transplantation (1 to 10 years post-transplant)
* Treatment with sirolimus + mycophenolate mofetil + steroids + ACE inhibitor or angiotensin II receptor antagonist + statin

Exclusion Criteria

* Treatment with a CNI or azathioprine
* Vascular rejection or biopsy-proven acute rejection within 3 months prior to screening
* Severe dyslipidemia Other protocol-defined inclusion / exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-02; Primary Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Renal function at M6 (glomerular filtration and tubular function).

SECONDARY OUTCOMES:
Renal function (other tubular function parameters)
Incidence of biopsy-proven acute rejections and CMV infections
Laboratory parameters: hemoglobin, WBC, T-cell sub-populations, platelets, transaminases, total cholesterol, HDL and LDL cholesterol, apolipoproteins A1 and B, triglycerides, fasting glucose, HbA1c, LH, FSH, testosterone and TSH
Mucous and cutaneous disorders
Adverse events and serious adverse events, premature study treatment discontinuations.
Monitoring of everolimus trough levels.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Novartis, Basel, Switzerland

REFERENCES:
- [Result] Kamar N, Jaafar A, Esposito L, Ribes D, Durand D, Di-Giambattista F, Tack I, Rostaing L. Conversion from sirolimus to everolimus in maintenance renal transplant recipients within a calcineurin inhibitor-free regimen: results of a 6-month pilot study. Clin Nephrol. 2008 Aug;70(2):118-25. doi: 10.5414/cnp70118. PMID 18793527